CLINICAL TRIAL: NCT04206332
Title: A Phase 1, Dose Escalation, Open-Label Clinical Trial With Experimental Controlled Human Malaria Infections (CHMI) to Evaluate Safety and Protective Efficacy of an Anti-Malaria Human Monoclonal Antibody, VRC-MALMAB0100-00-AB (CIS43LS), in Healthy, Malaria-Naive Adults
Brief Title: Trial to Evaluate CIS43LS in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 200017; 20-I-0017
Record Dates: First submitted 2019-12-19; First posted 2019-12-20 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Malaria
Keywords: Prevention and Control; Mosquito; Malaria Challenge; Parasitemia; Passive Immunization; Controlled Human Malaria Infection (CHMI)
MeSH Terms: conditions — Malaria; Parasitemia | interventions — CIS43LS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Part A, Group 1: CIS43LS (5 mg/kg IV) (Experimental): CIS43LS (5 mg/kg) administered by intravenous (IV) infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB
- Part A, Group 2: CIS43LS (5 mg/kg SC) (Experimental): CIS43LS (5 mg/kg) administered by subcutaneous (SC) injection (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB
- Part A, Group 3: CIS43LS (20 mg/kg IV) (Experimental): CIS43LS (20 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB
- Part A, Group 4A: CIS43LS (40 mg/kg IV) (Experimental): CIS43LS (40 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB
- Part A, Group 4B: CIS43LS (40 mg/kg IV) (Experimental): CIS43LS (40 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB
- Part A, Group 5: CHMI Controls (No Intervention): Control participants who did not receive CIS43LS and were enrolled to complete the controlled human malaria infection (CHMI); however, Group 5 did not undergo CHMI because of restrictions related to coronavirus disease 2019 (COVID-19)
- Part B, Group 6: CIS43LS (5 mg/kg SC) (Experimental): CIS43LS (5 mg/kg) administered by SC injection (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part B, Group 7: CIS43LS (20 mg/kg IV) (Experimental): CIS43LS (20 mg/kg) administered by IV infusion (Day 0)
  Part B, Group 7 participants included participants previously enrolled in Part A who received either 5 mg/kg IV (1), 5 mg/kg SC (1) or 20 mg/kg IV (2) in the first part of the study and newly enrolled Part B participants
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] (Other): Part B, Group 8 participants included participants previously enrolled in Part A who received CIS43LS (40 mg/kg IV) in the first part of the study but did not receive CIS43LS in Part B of the study. Group 8 participants were enrolled to complete the controlled human malaria infection (CHMI).
  Interventions: Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part B, Group 9: CIS43LS (40 mg/kg IV) (Experimental): CIS43LS (40 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part B, Group 10: CHMI Controls (Other): Control participants who did not receive CIS43LS and were enrolled to complete the controlled human malaria infection (CHMI)
  Interventions: Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part C, Group 11: CIS43LS (1 mg/kg IV) (Experimental): CIS43LS (1 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part C, Group 12: CIS43LS (5 mg/kg IV) (Experimental): CIS43LS (5 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part C, Group 13: CIS43LS (5 mg/kg SC) (Experimental): CIS43LS (5 mg/kg) administered by SC injection (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part C, Group 14: CIS43LS (10 mg/kg IV) (Experimental): CIS43LS (10 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part C, Group 15: CIS43LS (10 mg/kg SC) (Experimental): CIS43LS (10 mg/kg) administered by SC injection (Day 0)
  Interventions: Drug: VRC-MALMAB0100-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Part C, Group 16: CHMI Controls (Other): Control participants who did not receive CIS43LS and were enrolled to complete the controlled human malaria infection (CHMI)
  Interventions: Other: Plasmodium falciparum (P. falciparum) sporozoite challenge

INTERVENTIONS:
Drug: VRC-MALMAB0100-00-AB — VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein and incorporates an LS mutation to increase product half-life in plasma.
  Other Names: CIS43LS
  Arms: Part A, Group 1: CIS43LS (5 mg/kg IV); Part A, Group 2: CIS43LS (5 mg/kg SC); Part A, Group 3: CIS43LS (20 mg/kg IV); Part A, Group 4A: CIS43LS (40 mg/kg IV); Part A, Group 4B: CIS43LS (40 mg/kg IV); Part B, Group 6: CIS43LS (5 mg/kg SC); Part B, Group 7: CIS43LS (20 mg/kg IV); Part B, Group 9: CIS43LS (40 mg/kg IV); Part C, Group 11: CIS43LS (1 mg/kg IV); Part C, Group 12: CIS43LS (5 mg/kg IV); Part C, Group 13: CIS43LS (5 mg/kg SC); Part C, Group 14: CIS43LS (10 mg/kg IV); Part C, Group 15: CIS43LS (10 mg/kg SC)
Other: Plasmodium falciparum (P. falciparum) sporozoite challenge — Participants were exposed to bites on the forearm from Anopheles stephensi mosquitoes infected with P. falciparum (3D7 strain).
  Arms: Part B, Group 10: CHMI Controls; Part B, Group 6: CIS43LS (5 mg/kg SC); Part B, Group 7: CIS43LS (20 mg/kg IV); Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A]; Part B, Group 9: CIS43LS (40 mg/kg IV); Part C, Group 11: CIS43LS (1 mg/kg IV); Part C, Group 12: CIS43LS (5 mg/kg IV); Part C, Group 13: CIS43LS (5 mg/kg SC); Part C, Group 14: CIS43LS (10 mg/kg IV); Part C, Group 15: CIS43LS (10 mg/kg SC); Part C, Group 16: CHMI Controls

SUMMARY:
Background:

People get malaria when they are bitten by an infected mosquito. Malaria can be serious and sometimes deadly. Although there are medicines to treat malaria, there is no vaccine that fully prevents infection. Researchers want to test if an experimental drug can help.

Objective:

To test the safety and effectiveness of a drug called CIS43LS that could prevent malaria infection.

Eligibility:

Healthy people ages 18-50 who have never been infected with malaria

Design:

Participants were enrolled on the basis of eligibility criteria, evaluated by clinical laboratory tests, self-reported medical history, and physical examination.

Participants received CIS43LS either infused into a vein in their arm or injected into the fat under the skin. They were monitored for side effects for up to 4 hours after they received the drug. Participants received a thermometer and recorded their temperature and symptoms every day on/with/via a diary card for 7 days after administration. The administration site was checked for redness, swelling, itching or bruising.

Participants had up to 12 follow-up visits. At follow-up visits, participants had blood drawn and were checked for health changes or problems.

Most participants who received CIS43LS took part in a Controlled Human Malaria Infection Challenge (CHMI) along with control participants who did not receive CIS43LS. During the CHMI, mosquitoes carrying the malaria parasite bit participants in a controlled setting. The participants had clinic visits every day for up to 12 days starting 7 days after the CHMI. Participants were treated right away with antimalarial medication if they tested positive for malaria. Approximately 21 days after the CHMI, participants were treated with antimalarial medication for 3 days.

The study lasted 2-6 months depending on the participant's study group.

DETAILED DESCRIPTION:
This was a multicenter, three-part, first-in-human, Phase 1, open-label, dose escalation study to evaluate the dose, safety, tolerability and protective efficacy of an anti-malaria human monoclonal antibody, VRC-MALMAB0100-00-AB (CIS43LS). The primary objective was to evaluate the safety and tolerability of CIS43LS when administered by either intravenous (IV) or subcutaneous (SC) routes. The secondary objectives were to evaluate the pharmacokinetics of CIS43LS at each dose level, determine if IV or SC administration will confer protection following a controlled human malaria infection (CHMI), and estimate the lowest protective dose of CIS43LS.

Part A: Part A evaluated the doses and routes in an open-label, dose escalation design.

Part B: Part B evaluated CIS43LS doses and routes prior to CHMI in participants previously enrolled in Part A and new Part B enrollees. A subgroup of participants from Part A continued to Part B, and some received a second CIS43LS dose intravenously. Additional participants were enrolled in Part B and received CIS43LS intravenously.

Part C: Part C evaluated CIS43LS doses and routes needed to reach a threshold of protection by assessing serum concentration prior to CHMI in a dose down design.

Study Product:

CIS43LS is a human immunoglobulin gamma-1 (IgG1) monoclonal antibody that was developed and manufactured by the National Institutes of Health (NIH) Vaccine Research Center (VRC). A recombinant Chinese hamster ovary DG44 clonal cell line14 developed by the Vaccine Production Program was transferred to the VRC pilot plant for clinical material manufacture. The study product was manufactured according to Good Manufacturing Practice at the VRC pilot plant operated by the Vaccine Clinical Materials Program, Leidos Biomedical Research (Frederick, MD, USA).

VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein and incorporates an LS mutation to increase product half-life in plasma.

Participants:

A total of 71 participants enrolled in the study as follows:

Part A: 29 participants enrolled in Groups 1-5

Part B: 21* participants enrolled in Groups 6-10

*Out of the 21 Part B participants, 11 were newly enrolled and 10 were Part A participants who re-enrolled.

Of the 10 Part A participants who re-enrolled in Part B, 3 were back up participants who did not receive additional CIS43LS or CHMI and were terminated early because they were not needed.

Therefore, only 18 participants were actively enrolled in Part B: 11 newly enrolled and 7 Part A participants who re-enrolled.

Part C: 31 participants enrolled in Groups 11-16

Of the 71 participants enrolled, 47 participants received at least one dose of CIS43LS and 43 participants completed the CHMI.

Of the 47 participants who received CIS43LS, 4 participants who received a dose in Part A were also enrolled in Part B and received a second dose as follows:

* one participant received a 5 mg/kg IV dose in Part A and 20 mg/kg IV dose in Part B,
* one participant received a 5 mg/kg SC dose in Part A and 20 mg/kg IV dose in Part B, and
* two participants received a 20 mg/kg IV dose in Part A and Part B.

Therefore, a total of 51 doses of CIS43LS were administered to 47 participants as follows:

* 7 doses of 1 mg/kg IV
* 8 doses of 5 mg/kg SC
* 8 doses of 5 mg/kg IV
* 3 doses of 10 mg/kg IV
* 4 doses of 10 mg/kg SC
* 9 doses of 20 mg/kg IV and
* 12 doses of 40 mg/kg IV

Study Duration:

Participants who received CIS43LS were followed for up to 24 weeks after product administration. Control participants were followed through 7 weeks after CHMI.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Able and willing to complete the informed consent process
  2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
  3. Available for clinical follow-up through the last study visit
  4. 18 to 50 years of age
  5. In good general health without clinically significant medical history
  6. Physical examination without clinically significant findings within the 56 days prior to enrollment
  7. Weight <= 115 kg (for all groups except Groups 5, 10, and 16) and < 100 kg for Group 15
  8. Adequate venous access if assigned to an IV group or adequate subcutaneous tissue if assigned to an SC group
  9. Willing to have blood samples collected, stored indefinitely, and used for research purposes
  10. Agrees to participate in a controlled human malaria infection (CHMI) and to comply with post-CHMI follow-up requirements (except Group 4B)
  11. Agrees to refrain from blood donation to blood banks for 3 years following participation in CHMI (except Group 4B)
  12. Agrees not to travel to a malaria endemic region during the entire course of study participation

      Laboratory Criteria within 56 days prior to enrollment:
  13. White Blood Cell (WBC) 2,500-12,000/mm^3
  14. WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval
  15. Platelets = 125,000 - 500,000/mm^3
  16. Hemoglobin within institutional normal range or accompanied by the PI or designee approval
  17. Creatinine <= 1.1 x upper limit of normal (ULN)
  18. Alanine aminotransferase (ALT) <= 1.25 x ULN
  19. Negative for HIV infection by an FDA approved method of detection

      Laboratory Criteria documented any time prior to enrollment:
  20. Negative sickle cell screening test
  21. Negative troponin test (except Group 4B)
  22. Electrocardiogram (ECG) without clinically significant abnormalities (examples may include: pathologic Q waves, significant ST-T wave changes, left ventricular hypertrophy, any non-sinus rhythm excluding isolated premature atrial contractions, right or left bundle branch block, advanced A-V heart block). ECG abnormalities determined by a cardiologist to be clinically insignificant as related to study participation do not preclude study enrollment (except Group 4B)
  23. No evidence of increased cardiovascular disease risk; defined as >10% five-year risk by the non-laboratory method (except Group 4B)

      Criteria Specific to Women:
  24. Postmenopausal for at least 1 year, post-hysterectomy or bilateral oophorectomy, or if of childbearing potential:

      1. Negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on day of enrollment, and prior to product administration and CHMI, and
      2. Agrees to use an effective means of birth control through the duration of study participation
* EXCLUSION CRITERIA:

  1. Woman who is breast-feeding or planning to become pregnant during study participation
  2. Previous receipt of a malaria vaccine
  3. History of malaria infection
  4. History of severe infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) defined per FDA guidance
  5. Active SARS-CoV-2 infection
  6. Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the study
  7. Hypertension that is not well controlled
  8. Receipt of any investigational study product within 28 days prior to enrollment (note: Emergency Use Authorization Coronavirus Disease 2019 (COVID-19) vaccine is not exclusionary)
  9. Receipt of any live attenuated vaccines within 28 days prior to enrollment
  10. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular injections or blood draws
  11. History of a splenectomy, sickle cell disease or sickle cell trait
  12. History of skeeter syndrome or anaphylactic response to mosquito-bites (except Group 4B)
  13. Known intolerance to chloroquine phosphate, atovaquone or proguanil (except Group 4B)
  14. Use or planned use of any drug, including antibiotics, with antimalarial activity within 4 weeks prior to CHMI
  15. History of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine (except Group 4B)
  16. Anticipated use of medications known to cause drug reactions with chloroquine or atovaquone-proguanil (Malarone) such as cimetidine, metoclopramide, antacids, and kaolin (except Group 4B)
  17. Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer, including but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Program Leadership:ctpleadership@mail.nih.gov, Study Director — VRC, National Institute of Allergy and Infectious Diseases, National Institutes of Health
Locations (2):
- United States (2):
  - University of Maryland Baltimore, Center for Vaccine Development, Baltimore, Maryland
  - VRC Clinic, NIH Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not shared because it has limited value in a small phase 1 trial of healthy volunteers. We instead report non-IPD data as required in ClinicalTrials.gov.

REFERENCES:
- [Background] Gaudinski MR, Coates EE, Novik L, Widge A, Houser KV, Burch E, Holman LA, Gordon IJ, Chen GL, Carter C, Nason M, Sitar S, Yamshchikov G, Berkowitz N, Andrews C, Vazquez S, Laurencot C, Misasi J, Arnold F, Carlton K, Lawlor H, Gall J, Bailer RT, McDermott A, Capparelli E, Koup RA, Mascola JR, Graham BS, Sullivan NJ, Ledgerwood JE; VRC 608 Study team. Safety, tolerability, pharmacokinetics, and immunogenicity of the therapeutic monoclonal antibody mAb114 targeting Ebola virus glycoprotein (VRC 608): an open-label phase 1 study. Lancet. 2019 Mar 2;393(10174):889-898. doi: 10.1016/S0140-6736(19)30036-4. Epub 2019 Jan 24. PMID 30686586
- [Background] Ishizuka AS, Lyke KE, DeZure A, Berry AA, Richie TL, Mendoza FH, Enama ME, Gordon IJ, Chang LJ, Sarwar UN, Zephir KL, Holman LA, James ER, Billingsley PF, Gunasekera A, Chakravarty S, Manoj A, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, K C N, Murshedkar T, DeCederfelt H, Plummer SH, Hendel CS, Novik L, Costner PJ, Saunders JG, Laurens MB, Plowe CV, Flynn B, Whalen WR, Todd JP, Noor J, Rao S, Sierra-Davidson K, Lynn GM, Epstein JE, Kemp MA, Fahle GA, Mikolajczak SA, Fishbaugher M, Sack BK, Kappe SH, Davidson SA, Garver LS, Bjorkstrom NK, Nason MC, Graham BS, Roederer M, Sim BK, Hoffman SL, Ledgerwood JE, Seder RA. Protection against malaria at 1 year and immune correlates following PfSPZ vaccination. Nat Med. 2016 Jun;22(6):614-23. doi: 10.1038/nm.4110. Epub 2016 May 9. PMID 27158907
- [Background] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949
- [Background] Kayentao K, Ongoiba A, Preston AC, Healy SA, Doumbo S, Doumtabe D, Traore A, Traore H, Djiguiba A, Li S, Peterson ME, Telscher S, Idris AH, Kisalu NK, Carlton K, Serebryannyy L, Narpala S, McDermott AB, Gaudinski M, Traore S, Cisse H, Keita M, Skinner J, Hu Z, Zeguime A, Ouattara A, Doucoure M, Dolo A, Djimde A, Traore B, Seder RA, Crompton PD; Mali Malaria mAb Trial Team. Safety and Efficacy of a Monoclonal Antibody against Malaria in Mali. N Engl J Med. 2022 Nov 17;387(20):1833-1842. doi: 10.1056/NEJMoa2206966. Epub 2022 Oct 31. PMID 36317783
- [Result] Gaudinski MR, Berkowitz NM, Idris AH, Coates EE, Holman LA, Mendoza F, Gordon IJ, Plummer SH, Trofymenko O, Hu Z, Campos Chagas A, O'Connell S, Basappa M, Douek N, Narpala SR, Barry CR, Widge AT, Hicks R, Awan SF, Wu RL, Hickman S, Wycuff D, Stein JA, Case C, Evans BP, Carlton K, Gall JG, Vazquez S, Flach B, Chen GL, Francica JR, Flynn BJ, Kisalu NK, Capparelli EV, McDermott A, Mascola JR, Ledgerwood JE, Seder RA; VRC 612 Study Team. A Monoclonal Antibody for Malaria Prevention. N Engl J Med. 2021 Aug 26;385(9):803-814. doi: 10.1056/NEJMoa2034031. Epub 2021 Aug 11. PMID 34379916
- [Result] Lyke KE, Berry AA, Mason K, Idris AH, O'Callahan M, Happe M, Strom L, Berkowitz NM, Guech M, Hu Z, Castro M, Basappa M, Wang L, Low K, Holman LA, Mendoza F, Gordon IJ, Plummer SH, Trofymenko O, Strauss KS, Joshi S, Shrestha B, Adams M, Chagas AC, Murphy JR, Stein J, Hickman S, McDougal A, Lin B, Narpala SR, Vazquez S, Serebryannyy L, McDermott A, Gaudinski MR, Capparelli EV, Coates EE, Wu RL, Ledgerwood JE, Dropulic LK, Seder RA; VRC 612 Part C Study Team. Low-dose intravenous and subcutaneous CIS43LS monoclonal antibody for protection against malaria (VRC 612 Part C): a phase 1, adaptive trial. Lancet Infect Dis. 2023 May;23(5):578-588. doi: 10.1016/S1473-3099(22)00793-9. Epub 2023 Jan 25. PMID 36708738
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0017.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited for Parts A and B of the study at the NIH Clinical Center in Bethesda, Maryland, USA. Healthy adults were recruited for Part C of the study at the University of Maryland, Baltimore Center for Vaccine Development and Global Health, Baltimore, MD, USA.
Pre-assignment Details: A subgroup of 10 participants from Part A who continued to Part B is counted twice: 4 Part A participants received a 2nd CIS43LS dose of 20 mg/kg IV in Part B (1 received 5 mg/kg IV, 1 received 5 mg/kg SC, and 2 received 20 mg/kg IV in Part A) and 6 did not receive CIS43LS in Part B: 3 enrolled as back up in the 20 mg/kg IV group (1 received 5 mg/kg IV, 1 received 5 mg/kg SC and 1 received 20 mg/kg IV in Part A) and 3 enrolled in CHMI (2 received 40 mg/kg IV and 1 enrolled in CHMI in Part A)
Groups:
- Part B, Group 7: CIS43LS (20 mg/kg IV): CIS43LS (20 mg/kg) administered by IV infusion (Day 0)
  Part B, Group 7 participants included participants previously enrolled in Part A who received either 5 mg/kg IV (1), 5 mg/kg SC (1) or 20 mg/kg IV (2) in the first part of the study and newly enrolled Part B participants
  VRC-MALMAB0100-00-AB: VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein and incorporates an LS mutation to increase product half-life in plasma.
  Plasmodium falciparum (P. falciparum) sporozoite challenge: Participants were exposed to bites on the forearm from Anopheles stephensi mosquitoes infected with P. falciparum (3D7 strain).
Period: Part A
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part A, Group 5: CHMI Controls | Part B, Group 6: CIS43LS (5 mg/kg SC) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part B, Group 10: CHMI Controls | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC) | Part C, Group 16: CHMI Controls
Started | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Product Administration | 4 | 4 | 5 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Controlled Human Malaria Infection (CHMI) | 0 (CHMI canceled because of restrictions related to coronavirus disease 2019 (COVID-19)) | 0 (CHMI canceled because of restrictions related to coronavirus disease 2019 (COVID-19)) | 0 (CHMI canceled because of restrictions related to coronavirus disease 2019 (COVID-19)) | 0 (CHMI canceled because of restrictions related to coronavirus disease 2019 (COVID-19)) | 0 (CHMI canceled because of restrictions related to coronavirus disease 2019 (COVID-19)) | 0 (CHMI canceled because of restrictions related to coronavirus disease 2019 (COVID-19)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 3 | 5 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — CHMI canceled because of restrictions related to coronavirus disease 2019 (COVID-19) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part A, Group 5: CHMI Controls | Part B, Group 6: CIS43LS (5 mg/kg SC) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part B, Group 10: CHMI Controls | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC) | Part C, Group 16: CHMI Controls
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 (Seven (7) participants from Part A enrolled in Part B, Group 7: CIS43LS (20 mg/kg IV). Of the 7 participants who enrolled in Part B, only 4 received a second product administration.) | 2 (Two (2) participants from Part A enrolled in Part B, Group 8: CHMI.) | 4 | 8 (One (1) participant from Part A enrolled in Part B, Group 10: CHMI.) | 0 | 0 | 0 | 0 | 0 | 0
Received Product Administration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Controlled Human Malaria Infection (CHMI) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Back up participants who did not receive CIS43LS or CHMI because they were not needed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part A, Group 5: CHMI Controls | Part B, Group 6: CIS43LS (5 mg/kg SC) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part B, Group 10: CHMI Controls | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC) | Part C, Group 16: CHMI Controls
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 4 | 4 | 8
Received Product Administration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 3 (One participant enrolled, but product not given: Withdrew consent on day of planned administration) | 4 | 0
Completed Controlled Human Malaria Infection (CHMI) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 3 | 4 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 2 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Not completed — Back up participants who did not receive CIS43LS or CHMI because they were not needed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 71 participants enrolled; however, 10 participants previously enrolled in Part A and who were later enrolled in Part B are counted twice (once in Part A and again in Part B).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part A, Group 5: CHMI Controls | Part B, Group 6: CIS43LS (5 mg/kg SC) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part B, Group 10: CHMI Controls | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC) | Part C, Group 16: CHMI Controls | Total
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 7 | 2 | 4 | 8 | 7 | 4 | 4 | 4 | 4 | 8 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Each row population reports Baseline Characteristics data separately for each part of the study (e.g., "Part A", "Part B", and "Part C").
  years
    Part A: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
    Part A | 26.5 (5.1) | 23.5 (3.7) | 29.4 (5.4) | 35.0 (10.2) | 25.3 (4.0) | 30.5 (8.9) |  |  |  |  |  |  |  |  |  |  |  | 29.0 (7.6)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Part B |  |  |  |  |  |  |  | 25.1 (4.2) | 31.5 (10.6) | 26.8 (3.4) | 30.1 (4.5) |  |  |  |  |  |  | 28.0 (5.1)
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 4 | 4 | 8 | 31
    Part C |  |  |  |  |  |  |  |  |  |  |  | 38.6 (8.7) | 30.5 (5.6) | 37.3 (7.4) | 31.0 (7.6) | 28.3 (3.3) | 32.5 (9.7) | 33.5 (8.1)
Age, Customized [Count of Participants; unit: Participants] — Population: Each row population reports Baseline Characteristics data separately for each part of the study (e.g., "Part A", "Part B", and "Part C").
  Participants
    Part A: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
    Part A: 18-20 years | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Part A: 21-30 years | 3 | 4 | 3 | 2 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
    Part A: 31-40 years | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
    Part A: 41-50 years | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Part B: 18-20 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Part B: 21-30 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Part B: 31-40 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 5
    Part B: 41-50 years | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 4 | 4 | 8 | 31
    Part C: 18-20 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Part C: 21-30 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 4 | 12
    Part C: 31-40 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 2 | 11
    Part C: 41-50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each row population reports Baseline Characteristics data separately for each part of the study (e.g., "Part A", "Part B", and "Part C").
  Participants
    Part A: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
    Part A: Female | 2 | 2 | 1 | 4 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17
    Part A: Male | 2 | 2 | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Part B: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 11
    Part B: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 4 | 4 | 8 | 31
    Part C: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 4 | 3 | 4 | 18
    Part C: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 0 | 1 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row population reports Baseline Characteristics data separately for each part of the study (e.g., "Part A", "Part B", and "Part C").
  Participants
    Part A: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
    Part A: Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    Part A: Not Hispanic or Latino | 3 | 4 | 4 | 5 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26
    Part A: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Part B: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Part B: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 19
    Part B: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 4 | 4 | 8 | 31
    Part C: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Part C: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 3 | 4 | 8 | 30
    Part C: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Each row population reports Baseline Characteristics data separately for each part of the study (e.g., "Part A", "Part B", and "Part C").
  Participants
    Part A: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
    Part A: Asian | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
    Part A: Black or African American | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Part A: White | 4 | 1 | 3 | 4 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Part A: Multiracial | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Part B: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7
    Part B: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Part B: White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 9
    Part B: Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 4 | 4 | 8 | 31
    Part C: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part C: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 6
    Part C: White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 2 | 2 | 4 | 7 | 24
    Part C: Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight (kg) [Mean (Standard Deviation); unit: kg] — Weight was collected at enrollment day per the protocol Schedule of Evaluations (SoE) for each group. The weight measurement for the Part C, Group 16 CHMI control participants represents weight collected during screening in the screening protocol as the protocol SoE did not require weight collection at enrollment for Group 16. Therefore, the overall weight calculation for Part C does not include the Group 16 participants as noted in the Measure Analysis Population Description below. Population: Each row population reports baseline characteristics data separately for each part of the study. Part C: A total of 22 weights were collected at enrollment and included in the overall weight measurement: one Group 14 participant withdrew prior to product administration and weight collection, and 8 Group 16 participants had weight collected during screening but not at enrollment. Weight collected for Group 16 participants in the screening protocol is excluded from the overall weight evaluation.
  kg
    Part A: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
    Part A | 67.1 (8.8) | 70.5 (15.1) | 74.4 (14.7) | 73.8 (12.7) | 66.2 (19.5) | 66.9 (14.8) |  |  |  |  |  |  |  |  |  |  |  | 69.8 (13.4)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Part B |  |  |  |  |  |  |  | 65.0 (13.4) | 72.1 (1.3) | 75.9 (13.5) | 74.9 (16.0) |  |  |  |  |  |  | 71.1 (13.8)
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 3 | 4 | 8 | 30
    Part C |  |  |  |  |  |  |  |  |  |  |  | 75.6 (18.9) | 70.8 (3.2) | 85.5 (14.5) | 66.6 (4.1) | 74.6 (19.5) | 70.8 (14.0) | 75.1 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of CIS43LS Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after CIS43LS product administration, at approximately Week 1
Population: Population included all enrolled participants who received CIS43LS and provided safety data (via diary card). A subgroup of 4 participants from Part A who continued to Part B are counted twice, and received a second CIS43LS dose intravenously (IV): 4 received CIS43LS at a dose of 20 mg/kg IV in Part B (1 had previously received 5 mg/kg IV, 1 had received 5 mg/kg subcutaneously, and 2 had received 20 mg/kg IV). No participants enrolled in Group 6: CIS43LS (5 mg/kg SC).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
Participants
  Pain/Tenderness: None | 4 | 1 | 5 | 3 | 3 | 2 | 4 | 4 | 4 | 4 | 3 | 3
  Pain/Tenderness: Mild | 0 | 3 | 0 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 1
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritis (Itching): None | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 3
  Pruritis (Itching): Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Pruritis (Itching): Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritis (Itching): Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 6 | 4 | 4 | 3 | 4
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: None | 4 | 4 | 5 | 4 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
  Bruising: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: Moderate | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 4 | 1 | 5 | 3 | 3 | 2 | 4 | 4 | 4 | 4 | 3 | 2
  Any Local Symptom: Mild | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 2
  Any Local Symptom: Moderate | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of CIS43LS Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after CIS43LS product administration, at approximately Week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
Participants
  Malaise: None | 4 | 4 | 5 | 4 | 3 | 2 | 4 | 6 | 3 | 3 | 2 | 3
  Malaise: Mild | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1
  Malaise: Moderate | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Aches: None | 4 | 2 | 4 | 3 | 3 | 4 | 4 | 6 | 3 | 4 | 3 | 3
  Muscle Aches: Mild | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Muscle Aches: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Muscle Aches: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 3 | 3 | 3 | 4 | 2 | 4 | 3 | 6 | 3 | 4 | 2 | 2
  Headache: Mild | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Headache: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
  Chills: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 3 | 4 | 5 | 5 | 3 | 3 | 4 | 5 | 4 | 4 | 3 | 4
  Nausea: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Nausea: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 4 | 4 | 5 | 4 | 3 | 4 | 4 | 7 | 3 | 4 | 3 | 3
  Joint Pain: Mild | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): None | 4 | 4 | 5 | 5 | 3 | 4 | 3 | 7 | 4 | 4 | 3 | 4
  Temperature (Fever): Mild | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 3 | 1 | 3 | 2 | 2 | 2 | 2 | 5 | 3 | 3 | 2 | 2
  Any Systemic Symptom: Mild | 0 | 3 | 2 | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 2
  Any Systemic Symptom: Moderate | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following CIS43LS Product Administration
Description: Unsolicited adverse event (AE) data collection included AEs of all severities from the date of product administration through the Day 28 post-product administration visit. At other time periods between study product administration and when greater than 4 weeks after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions that required ongoing medical management (reported as a separate outcome) were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after CIS43LS product administration
Population: Population included all enrolled participants who received CIS43LS and had safety data collected (via clinical assessment and/or lab results). A subgroup of 4 participants from Part A who continued to Part B are counted twice, and received a second CIS43LS dose intravenously (IV): 4 received CIS43LS at a dose of 20 mg/kg IV in Part B (1 had previously received 5 mg/kg IV, 1 received 5 mg/kg subcutaneously, and 2 received 20 mg/kg IV). No participants enrolled in Group 6: CIS43LS (5 mg/kg SC).
Measure: Count of Participants; unit: Participants
Groups:
- Part B, Group 7: CIS43LS (20 mg/kg IV): CIS43LS (20 mg/kg) administered by IV infusion (Day 0)
  Part B, Group 7 participants included participants previously enrolled in Part A who received either 5 mg/kg IV (1), 5 mg/kg SC (1) or 20 mg/kg IV (2) in the first part of the study and newly enrolled Part B participants
  VRC-MALMAB0100-00-AB: VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein. The monoclonal antibody was adapted resulting in an LS mutation found to increase product half-life in plasma.
  Plasmodium falciparum (P. falciparum) sporozoite challenge: Participants were exposed to bites on the forearm from Anopheles stephensi mosquitoes infected with P. falciparum (3D7 strain).
- Part B, Group 9: CIS43LS (40 mg/kg IV): CIS43LS (40 mg/kg) administered by IV infusion (Day 0)
  VRC-MALMAB0100-00-AB: VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein. The monoclonal antibody was adapted resulting in an LS mutation found to increase product half-life in plasma.
  Plasmodium falciparum (P. falciparum) sporozoite challenge: Participants were exposed to bites on the forearm from Anopheles stephensi mosquitoes infected with P. falciparum (3D7 strain).
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
Participants
  Related to Study Product | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
  Unrelated to Study Product | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 4
  Total Number of Participants who had One or More Non-Serious Unsolicited AE after CIS43LS | 4 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 2 | 2 | 4

4. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following Controlled Human Malaria Infection (CHMI)
Description: Unsolicited adverse event (AE) data collection included AEs of all severities from CHMI through the Day 28 post-CHMI visit. The relationship between an AE and CHMI was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after CHMI
Population: Population included all enrolled participants who completed CHMI and had safety data collected (via clinical assessment and/or laboratory results). Part A participants did not complete CHMI because of restrictions related to coronavirus disease 2019 (COVID-19). No participants enrolled in Part B, Group 6: CIS43LS (5 mg/kg SC).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part B, Group 10: CHMI Controls | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC) | Part C, Group 16: CHMI Controls
Number analyzed (Participants) | 4 | 2 | 3 | 6 | 7 | 4 | 4 | 3 | 4 | 6
Participants
  Related to CHMI | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Unrelated to CHMI | 1 | 0 | 0 | 1 | 3 | 2 | 3 | 2 | 3 | 0
  Total Number of Participants who had One or More Non-Serious Unsolicited AE after CHMI | 1 | 0 | 0 | 1 | 4 | 2 | 4 | 2 | 4 | 0

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following CIS43LS Product Administration
Description: SAEs were recorded from receipt of first study product administration through the last expected study visit at Week 24. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after CIS43LS product administration through the study participation, up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
Participants
  Related to Study Product | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Total number of Participants With SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following CIS43LS Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of first study product administration through the last expected study visit at Week 24. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after CIS43LS product administration through the study participation, up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following CIS43LS Product Administration
Description: Abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV) platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil counts) and chemistry (alanine aminotransferase (ALT) and creatinine). Complete Blood Count (CBC) with differential and Chemistry (ALT and creatinine) results were collected at different timepoints in Parts A, B and C throughout the study per the protocol's schedule of evaluations. Institutional laboratory normal ranges as well as the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 were used.
Time Frame: Day 0 through 4 weeks after CIS43LS product administration
Population: Population included all enrolled participants who received CIS43LS and had safety data collected via laboratory results. A subgroup of 4 participants from Part A who continued to Part B are counted twice, and received a second CIS43LS dose intravenously (IV): 4 received CIS43LS at a dose of 20 mg/kg IV in Part B (1 had previously received 5 mg/kg IV, 1 had received 5 mg/kg subcutaneously, and 2 had received 20 mg/kg IV). No participants enrolled in Group 6: CIS43LS (5 mg/kg SC).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 4 | 4 | 7 | 4 | 4 | 3 | 4
Participants
  Creatinine | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophil Count | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

8. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Maximum Observed Serum Concentration (Cmax) - (Part A and Part B)
Description: Serum concentrations of CIS43LS by dose group following a single administration. Cmax is the peak serum concentration that CIS43LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group. After subcutaneous injection, Cmax could not be fully calculated because of COVID-19-related interruptions in sample collection.
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: Population included all enrolled participants who received CIS43LS intravenously in Part A and/or Part B of the study with up to 24 weeks of pharmacokinetic data (N=25). The 5 mg/kg SC dose group could not be evaluated due to truncated sample collections. Data in the 20 mg/kg IV dose group included 1 who received 5 mg/kg IV, 1 who received 5 mg/kg SC, and 2 who received 20 mg/kg IV in Part A of the study and received a second dose of CIS43LS at 20 mg/kg of body weight in Part B of the study.
Measure: Mean (Standard Deviation); unit: μg/ml
Groups:
- Part A, Group 3 and Part B, Group 7: CIS43LS (20 mg/kg IV): CIS43LS (20 mg/kg) administered by IV infusion (Day 0)
  Part B, Group 7 participants included participants previously enrolled in Part A who received either 5 mg/kg IV (1), 5 mg/kg SC (1) or 20 mg/kg IV (2) in the first part of the study and newly enrolled Part B participants
  VRC-MALMAB0100-00-AB: VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein and incorporates an LS mutation to increase product half-life in plasma.
- Part A, Group 4A-4B and Part B, Group 9: CIS43LS (40 mg/kg IV): CIS43LS (40 mg/kg) administered by IV infusion (Day 0)
  VRC-MALMAB0100-00-AB: VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein and incorporates an LS mutation to increase product half-life in plasma.
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3 and Part B, Group 7: CIS43LS (20 mg/kg IV) | Part A, Group 4A-4B and Part B, Group 9: CIS43LS (40 mg/kg IV)
Number analyzed (Participants) | 4 | 0 | 9 | 12
μg/ml | 198.4 (28.2) |  | 934.6 (292.6) | 1764.4 (259.6)

9. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Maximum Observed Serum Concentration (Cmax) - (Part C)
Description: Serum concentrations of CIS43LS by dose group following a single administration. Cmax is the peak serum concentration that CIS43LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: Population included 22 enrolled participants who received CIS43LS: 21 CIS43LS participants with 24 weeks of pharmacokinetic data and one CIS43LS participant with 8 weeks of data (N=22). The participant with 8 weeks of data was assigned to the 10 mg/kg IV dose group and withdrew from the study at Day 15 post-CHMI.
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 7 | 4 | 4 | 3 | 4
μg/ml | 42.2 (10.4) | 223.5 (53.3) | 53.6 (8.5) | 383.7 (30.8) | 104 (19.2)

10. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Time to Reach Maximum Observed Serum Concentration (Tmax) - (Part A and Part B)
Description: Tmax is the time it takes to reach Cmax of CIS43LS after it has been administered; it is determined based on the summary PK curve for each dose group.
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Groups:
- Part A, Group 3 and Part B, Group 7: CIS43LS (20 mg/kg IV): CIS43LS (20 mg/kg) administered by IV infusion (Day 0)
  Part B, Group 7 participants included participants previously enrolled in Part A who received either 5 mg/kg IV (1), 5 mg/kg SC (1) or 20 mg/kg IV (2) in the first part of the study and newly enrolled Part B participants (4)
  VRC-MALMAB0100-00-AB: VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein and incorporates an LS mutation to increase product half-life in plasma.
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3 and Part B, Group 7: CIS43LS (20 mg/kg IV) | Part A, Group 4A-4B and Part B, Group 9: CIS43LS (40 mg/kg IV)
Number analyzed (Participants) | 4 | 0 | 9 | 12
days | 0.10 (0.08) |  | 0.07 (0.07) | 0.25 (0.5)

11. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Time to Reach Maximum Observed Serum Concentration (Tmax) - (Part C)
Description: as for outcome 10
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC)
Number analyzed (Participants) | 7 | 4 | 4 | 3 | 4
days | 0.02 (0) | 0.03 (0.02) | 14.32 (10.58) | 0.08 (0.09) | 16.6 (9.2)

12. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Beta Half-life (T1/2b) - (Part A and Part B)
Description: Beta half-life (T1/2b) is being reported for this study. Beta half-life (T1/2b) is the time required for half of the CIS43LS product to be eliminated from the serum. A two-compartmental population pharmacokinetic model with first order SC absorption was used to estimate overall beta half-life and bootstrap 90% confidence intervals (CIs).
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: Population included all enrolled participants who received CIS43LS subcutaneously and intravenously in Part A and/or Part B of the study with up to 24 weeks of pharmacokinetic. Due to pandemic related sample collection interruptions, Part A and Part B of the study were analyzed in conjunction to achieve adequate sample size for population pharmacokinetic model used to generate the population PK parameters as per protocol, including beta half-life and clearance.
Measure: Number (90% Confidence Interval); unit: days
Groups:
- Overall Part A and Part B CIS43LS Dose Groups: CIS43LS dose groups included adults who received CIS43LS (5 mg/kg SC, 5 mg/kg IV, 20 mg/kg IV, 40 mg/kg IV) intravenously or subcutaneously.
Arm/Group | Overall Part A and Part B CIS43LS Dose Groups
Number analyzed (Participants) | 29
days | 56 [51.9 to 77.0]

13. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Beta Half-life (T1/2b) - (Part C)
Description: Beta half-life (T1/2b) is the time required for half of the CIS43LS product to be eliminated from the serum. A two-compartmental population pharmacokinetic model with first order SC absorption was used to estimate overall beta half-life and bootstrap 95% confidence intervals (CIs).
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: Population included 22 enrolled participants who received CIS43LS: 21 CIS43LS participants with 24 weeks of pharmacokinetic (PK) data and one CIS43LS participant with 8 weeks of data (N=22). The participant with 8 weeks of data was assigned to the 10 mg/kg IV dose group and withdrew from the study at Day 15 post-CHMI. Per protocol, population PK analysis was performed to generate compartmental PK parameters, including clearance and half-life.
Measure: Number (95% Confidence Interval); unit: days
Groups:
- Overall Part C CIS43LS Dose Groups: CIS43LS dose groups included adults who received CIS43LS (1 mg/kg IV, 5 mg/kg SC, 5 mg/kg IV, 10 mg/kg SC, 10 mg/kg IV) intravenously or subcutaneously.
Arm/Group | Overall Part C CIS43LS Dose Groups
Number analyzed (Participants) | 22
days | 80 [76.5 to 83.2]

14. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Clearance Rate - (Part A and Part B)
Description: Rate of CIS43LS elimination divided by the plasma CIS43LS concentration; determined based on the summary pharmacokinetic (PK) curve for each study group. A two-compartmental population pharmacokinetic model with first order SC absorption was used to estimate overall clearance and bootstrap 90% confidence intervals (CIs).
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: Population included all enrolled participants who received CIS43LS subcutaneously and intravenously in Part A and/or Part B of the study with up to 24 weeks of pharmacokinetic (PK) data (N=29). Due to pandemic related sample collection interruptions, Part A and Part B of the study were analyzed in conjunction to achieve adequate sample size for population pharmacokinetic model used to generate the population PK parameters as per protocol, including beta half-life and clearance.
Measure: Number (90% Confidence Interval); unit: ml/day
Arm/Group | Overall Part A and Part B CIS43LS Dose Groups
Number analyzed (Participants) | 29
ml/day | 44.2 [39.6 to 47.9]

15. Secondary Outcome: Pharmacokinetic (PK) Parameters of CIS43LS: Clearance Rate - (Part C)
Description: Rate of CIS43LS elimination divided by the plasma CIS43LS concentration; determined based on the summary pharmacokinetic (PK) curve for each study group. A two-compartmental population pharmacokinetic model with first order SC absorption was used to estimate overall clearance and bootstrap 95% confidence intervals (CIs).
Time Frame: Baseline through 24 weeks after CIS43LS product administration
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: ml/day
Arm/Group | Overall Part C CIS43LS Dose Groups
Number analyzed (Participants) | 22
ml/day | 33.6 [30.7 to 36.5]

16. Secondary Outcome: Number of Participants Who Developed Plasmodium Falciparum (P. Falciparum) Parasitemia Following Controlled Human Malaria Infection (CHMI) Challenge (Part B)
Description: Parasitemia as determined by polymerase chain reaction (PCR) up to day 21 following CHMI to determine whether IV or SC administration of CIS43LS mediates protection against infectious P. falciparum following CHMI
Time Frame: Up to 21 days after CHMI
Population: Population included all participants in Part B who completed CHMI. Part A participants did not complete CHMI because of restrictions related to COVID-19. A subgroup of 4 study participants received 2 doses of CIS43LS: 1 received 5 mg/kg IV and 2 received 20 mg/kg in Part A of the study and received second antibody administration at 20 mg/kg IV in Part B of the study; 1 received 5 mg/kg SC in Part A and 20 mg/kg IV in Part B of the study. No participants enrolled in Group 6: CIS43LS (5 mg/kg SC).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part B, Group 10: CHMI Controls
Number analyzed (Participants) | 4 | 2 | 3 | 6
Participants | 0 | 0 | 0 | 5

17. Secondary Outcome: Number of Participants Who Developed Plasmodium Falciparum (P. Falciparum) Parasitemia Following Controlled Human Malaria Infection (CHMI) Challenge (Part C)
Description: Parasitemia as determined by polymerase chain reaction (PCR) up to day 21 following CHMI to determine the lowest dose of CIS43LS administered IV and SC that confers protection against infectious P. falciparum following CHMI in Part C of the study
Time Frame: Up to 21 days after CHMI
Population: Population included all participants in Part C who completed CHMI.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC) | Part C, Group 16: CHMI Controls
Number analyzed (Participants) | 7 | 4 | 4 | 3 | 4 | 6
Participants | 4 | 0 | 0 | 0 | 0 | 6

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data collection included AEs of all severities for the CIS43LS and/or CHMI recipients only. Unsolicited AEs were recorded from the date of investigational product (IP) administration through the Day 28 post-product administration visit and from CHMI through the Day 28 post-CHMI visit. After and between the indicated time periods, only serious AEs (SAEs) and new chronic medical conditions were recorded as AEs through the last expected study visit at Week 24.
Description: Solicited AEs collected through systematic assessment for IP recipients and unsolicited AEs collected for IP and/or CHMI recipients through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity. Counted twice: 10 in Part A who enrolled in Part B. Not counted: Group 6 and some in Groups 5 (n=8), 7 (n=3) and 14 (n=1) who received no IP/CHMI.
Groups:
- Part B, Group 7: CIS43LS (20 mg/kg IV): CIS43LS (20 mg/kg) administered by IV infusion (Day 0)
  Part B, Group 7 participants included participants previously enrolled in Part A who received either 5 mg/kg IV/SC or 20 mg/kg IV in the first part of the study and newly enrolled Part B participants
  VRC-MALMAB0100-00-AB: VRC-MALMAB0100-00-AB (CIS43LS) is a monoclonal antibody that recognizes a unique and conserved region of the Plasmodium falciparum (P. falciparum) circumsporozoite protein and incorporates an LS mutation to increase product half-life in plasma.
  Plasmodium falciparum (P. falciparum) sporozoite challenge: Participants were exposed to bites on the forearm from Anopheles stephensi mosquitoes infected with P. falciparum (3D7 strain).
Arm/Group | Part A, Group 1: CIS43LS (5 mg/kg IV) | Part A, Group 2: CIS43LS (5 mg/kg SC) | Part A, Group 3: CIS43LS (20 mg/kg IV) | Part A, Group 4A: CIS43LS (40 mg/kg IV) | Part A, Group 4B: CIS43LS (40 mg/kg IV) | Part B, Group 7: CIS43LS (20 mg/kg IV) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] | Part B, Group 9: CIS43LS (40 mg/kg IV) | Part B, Group 10: CHMI Controls | Part C, Group 11: CIS43LS (1 mg/kg IV) | Part C, Group 12: CIS43LS (5 mg/kg IV) | Part C, Group 13: CIS43LS (5 mg/kg SC) | Part C, Group 14: CIS43LS (10 mg/kg IV) | Part C, Group 15: CIS43LS (10 mg/kg SC) | Part C, Group 16: CHMI Controls
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/5 | 0/3 | 0/4 | 0/2 | 0/4 | 0/6 | 0/7 | 0/4 | 0/4 | 0/3 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/5 | 0/3 | 0/4 | 0/2 | 1/4 | 0/6 | 0/7 | 0/4 | 0/4 | 0/3 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 2/5 | 3/5 | 2/3 | 3/4 | 0/2 | 2/4 | 1/6 | 5/7 | 3/4 | 4/4 | 2/3 | 4/4 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Group 1: CIS43LS (5 mg/kg IV) (N=4) | Part A, Group 2: CIS43LS (5 mg/kg SC) (N=4) | Part A, Group 3: CIS43LS (20 mg/kg IV) (N=5) | Part A, Group 4A: CIS43LS (40 mg/kg IV) (N=5) | Part A, Group 4B: CIS43LS (40 mg/kg IV) (N=3) | Part B, Group 7: CIS43LS (20 mg/kg IV) (N=4) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] (N=2) | Part B, Group 9: CIS43LS (40 mg/kg IV) (N=4) | Part B, Group 10: CHMI Controls (N=6) | Part C, Group 11: CIS43LS (1 mg/kg IV) (N=7) | Part C, Group 12: CIS43LS (5 mg/kg IV) (N=4) | Part C, Group 13: CIS43LS (5 mg/kg SC) (N=4) | Part C, Group 14: CIS43LS (10 mg/kg IV) (N=3) | Part C, Group 15: CIS43LS (10 mg/kg SC) (N=4) | Part C, Group 16: CHMI Controls (N=6)
Perirectal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Group 1: CIS43LS (5 mg/kg IV) (N=4) | Part A, Group 2: CIS43LS (5 mg/kg SC) (N=4) | Part A, Group 3: CIS43LS (20 mg/kg IV) (N=5) | Part A, Group 4A: CIS43LS (40 mg/kg IV) (N=5) | Part A, Group 4B: CIS43LS (40 mg/kg IV) (N=3) | Part B, Group 7: CIS43LS (20 mg/kg IV) (N=4) | Part B, Group 8: CHMI [CIS43LS (40 mg/kg IV) in Part A] (N=2) | Part B, Group 9: CIS43LS (40 mg/kg IV) (N=4) | Part B, Group 10: CHMI Controls (N=6) | Part C, Group 11: CIS43LS (1 mg/kg IV) (N=7) | Part C, Group 12: CIS43LS (5 mg/kg IV) (N=4) | Part C, Group 13: CIS43LS (5 mg/kg SC) (N=4) | Part C, Group 14: CIS43LS (10 mg/kg IV) (N=3) | Part C, Group 15: CIS43LS (10 mg/kg SC) (N=4) | Part C, Group 16: CHMI Controls (N=6)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Administration site pain (General disorders) | 0 | 3 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Administration site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Administration site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Administration site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04206332/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT04206332/ICF_000.pdf